CLINICAL TRIAL: NCT02007538
Title: Assessment of Adequacy and Characteristics Molecular of the Sample Obtained by Fine-needle Aspiration (FNA) Cytology Lung, Mounted With Thin Prep Compared to the Conventional Smear, in the Diagnosis of Lung Cancer.
Brief Title: Thin Prep Versus Traditional Cytological Procedure for Lung Cancer
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Papi, MD, professor in respiratory medicine, Università degli Studi di Ferrara
Other Study IDs: FR01
Record Dates: First submitted 2013-05-22; First posted 2013-12-11 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Bronchoscopy; Fine Need Aspiration; Cytochemical Assays
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thin Prep: Samples obtained from this group will be tested with thin prep
- Control Group: Samples obtained from this group will be tested with conventional procedure.

SUMMARY:
In the diagnosis of lung cancer, the cytological sample obtained during Bronchoscopy (FBS), has an increasingly important role in the characterization of malignancy. The cytological sample can be harvested during bronchoscopy by bronchial brushing, bronchial lavages or fine needle aspiration. Immunocytochemical staining allows not only to discriminate between small cell lung cancer versus non-small cell lung cancer (NSCLC), but also to identify the expression of specific markers such as TTF-1, CK7, CK20, 4A4, 34βE12 and p63. Thin Prep is a technique for cytological assay already validated and largely used in the immunocytochemical determination of gynaecologic specimens. Further Studies are required to asses the accuracy of this technique compared to conventional smear in cytological airway samples obtained by fine needle aspiration.

DETAILED DESCRIPTION:
Patients undergoing FBS for lung cancer diagnosis purpose will be enrolled in the study. During FBS Fine Need Aspiration (FNA) will be performed. Four samplings by FNA will be performed in each patient. Two samplings will be processed with thin prep technique and two samplings with the traditional procedure. To avoid sampling procedures-related bias, the first harvested sample will be randomly tested with Thin Prep or Traditional technique.

ELIGIBILITY:
Inclusion Criteria:

* FBS undergoing bronchoscopy for diagnostic purpose of lung cancer.
* Informed consent.
* ASA Classification 1-3.

Exclusion Criteria:

* Patients intubated.
* Patients with respiratory failure.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected lung cancer
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
total cell counts | the participants will be sampled at the time of recruitment (i.e. the day of the bronchoscopy) and they will be followed until the definitive histological diagnosis, an expected average of 8 weeks
  To compare the recovered total cell counts in the samples processed by thin prep technique Vs conventional procedure

SECONDARY OUTCOMES:
Marker Expression | the participants will be sampled at the time of recruitment (i.e. the day of the bronchoscopy) and they will be followed until the definitive histological diagnosis, an expected average of 8 weeks
  to evaluate the expression of a pannel of markers evaluated by immonocytochemistry in samples processed with thin prep procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Papi, MD, Principal Investigator — Azienda Ospedaliera Universitaria di Ferrara
Locations (1):
- Bronchoscopy Unit, Section of Repiratory Disease, azienda ospedaliera universitaria di Ferrara, Ferrara, Italy